CLINICAL TRIAL: NCT00291928
Title: A Double-blind, Randomized, Placebo Controlled, Dose Escalation, Multi-centerphase I/II Trial of HuMax-CD20, a Fully Human Monoclonal Anti-CD20antibody, in Patients With Active Rheumatoid Arthritis Who Have Previously Failedone or More Disease Modifying Anti-rheumatic Drugs
Brief Title: HuMax-CD20 in Active Rheumatoid Arthritis, Phase I/II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 112657; HX-CD20-403 (Other: GENMAB)
Record Dates: First submitted 2006-02-14; First posted 2006-02-15 (Estimated); Last update posted 2012-11-12 (Estimated); Status verified 2012-11

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Medicare Part B

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dose ranging (Placebo Comparator): A double-blind, placebo controlled, dose escalation part randomized within each of 3 sequential cohorts (Part A),
  Interventions: Drug: Part A
- Parallel Arm RCT (Placebo Comparator): a parallel group part with randomization into one of 4 treatment arms (Part B).
  Interventions: Drug: Part B

INTERVENTIONS:
Drug: Part A — Part A Cohort 1: HuMax-CD20 300 mg at Days 0 and 14 or Placebo at Days 0 and 14 Cohort 2: HuMax-CD20 700 mg at Days 0 and 14 or Placebo at Days 0 and 14 Cohort 3: HuMax-CD20 1000 mg at Days 0 and 14 or Placebo at Days 0 and 14
  Arms: Dose ranging
Drug: Part B — Part B Group 1: HuMax-CD20 300 mg at Days 0 and 14 Group 2: HuMax-CD20 700 mg at Days 0 and 14 Group 3: HuMax-CD20 1000 mg at Days 0 and 14 Group 4: Placebo at Days 0 and 14
  Arms: Parallel Arm RCT

SUMMARY:
The purpose of this trial is primarily to investigate the safety profile of HuMax-CD20 in patients with active RA. Furthermore, the trial is designed to identify the dose levels to be used in future trials (based on evaluations of safety, pharmacokinetics and ACR and DAS responses).

DETAILED DESCRIPTION:
This trial consists of a double-blind, placebo controlled, dose escalation part with randomization to trial treatment within each of three sequential cohorts (Part A), and a parallel group part with randomization into one of four treatment arms (Part B). Patients in Parts A and B will receive two infusions of either HuMax-CD20 (300 mg, 700 mg, or 1000 mg) or placebo and will be followed for safety, efficacy, and pharmacokinetic measurements for 24 weeks. Hereafter patients will be followed every 12 weeks until B-cells (CD19+ cells) have returned to baseline levels. For patients in Part B, the follow-up visits at 36 and 48 weeks after initial trial treatment (Follow-up Visits 1 and 2) will include additional measurements of safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Active rheumatoid arthritis according to the American College of Rheumatology of at least six months duration with six or more swollen and six or more tender joints (of 28 joints) and Erythrocyte Sedimentation Rate (ESR) ≥ 22 mm/h and/or C-Reactive Protein (CRP) ≥ 10 mg/L (1 mg/dL).
* Treatment failure to one or more DMARDs.
* Treatment with methotrexate (7.5-25 mg/wk) for at least 12 weeks and at a stable dose for at least 4 weeks prior to planned start of trial treatment.

Exclusion Criteria:

* Use of DMARDs other than methotrexate.
* Current or previous (within four weeks of screening) participation in any other clinical trial.
* Previous exposure to other biological products within 4 weeks prior to planned start of trial treatment, and/or exposure to anti-CD20 antibodies within two years before screening for this trial.
* Any use of cyclophosphamide, nitrogen mustard, chlorambucil or other alkylating agents within five years before screening for this trial.
* Active autoimmune disease (other than RA and RA-associated secondary diseases) requiring immunosuppressive therapy.
* Past or current malignancy, except for resected cervical carcinoma Stage 1B or less, non-invasive basal cell and squamous cell skin carcinoma, malignant melanoma with a complete response of a duration of > 10 years, or other cancer diagnoses with a complete response of a duration of > 5 years.
* Chronic or current infectious disease including known or suspected positive serology for HIV, hepatitis B, or hepatitis C.
* Clinically significant cardiac disease, or history of significant cerebrovascular disease.
* Significant concurrent, uncontrolled medical condition including, but not limited to: renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, neurological, cerebral, or psychiatric disease.
* Breast feeding women, women with a positive pregnancy test at screening, or women of childbearing potential not willing to use adequate contraception during the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2005-02; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of HuMax-CD20 in patients with active rheumatoid arthritis | 24 weeks
To evaluate the efficacy of HuMax-CD20 in patients with active rheumatoid arthritis using the American College of Rheumatology (ACR) Response Assessment and Disease Activity Score (DAS) at 12 to 24 weeks after initiation of treatment | 24 weeks

SECONDARY OUTCOMES:
To evaluate the efficacy of HuMax-CD20 in patients with active rheumatoid arthritis by measuring the degree and duration of B-cell depletion | 24 weeks
To determine the pharmacokinetic profile of HuMax-CD20 in patients with active rheumatoid arthritis | 24 weeks
To determine host immune response, Human Anti Human Antibodies (HAHA), against HuMax-CD20 | 24 weeks
To evaluate the efficacy of HuMax-CD20 in patients with active rheumatoid arthritis using the American College of Rheumatology (ACR) Response Assessment and Disease Activity Score (DAS) at 36 & 48 weeks after initiation of treatment | 48 weeks
To evaluate if Fc-receptor polymorphism influences the safety and efficacy of HuMax-CD20 in patients with active rheumatoid arthritis | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Derived] Struemper H, Sale M, Patel BR, Ostergaard M, Osterborg A, Wierda WG, Hagenbeek A, Coiffier B, Jewell RC. Population pharmacokinetics of ofatumumab in patients with chronic lymphocytic leukemia, follicular lymphoma, and rheumatoid arthritis. J Clin Pharmacol. 2014 Jul;54(7):818-27. doi: 10.1002/jcph.268. Epub 2014 Jan 28. PMID 24443277
- [Derived] Ostergaard M, Baslund B, Rigby W, Rojkovich B, Jorgensen C, Dawes PT, Wiell C, Wallace DJ, Tamer SC, Kastberg H, Petersen J, Sierakowski S. Ofatumumab, a human anti-CD20 monoclonal antibody, for treatment of rheumatoid arthritis with an inadequate response to one or more disease-modifying antirheumatic drugs: results of a randomized, double-blind, placebo-controlled, phase I/II study. Arthritis Rheum. 2010 Aug;62(8):2227-38. doi: 10.1002/art.27524. PMID 20506254